CLINICAL TRIAL: NCT04295733
Title: Evaluation of Safety, Tolerability and Immunogenicity of Two Doses of the 4CMenB Vaccine in Adults With an Immunodeficiency
Brief Title: Safety, Tolerability and Immunogenicity of 4CMenB Vaccine(2 Doses) in Adults With an Immunodeficiency
Acronym: 4CMenB
Status: Completed | Type: Observational
Sponsor: Ospedale Policlinico San Martino (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Laura Sticchi, Principal Investigator, Ospedale Policlinico San Martino
Other Study IDs: 4CMenB
Record Dates: First submitted 2020-02-24; First posted 2020-03-04 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Acquired Immunodeficiency
MeSH Terms: interventions — 4CMenB vaccine; Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (3):
- Cohort 1: Hematopoietic Stem Celi Transplant (HSCT) patients
  Interventions: Biological: 4CMenB (Bexsero®) vaccine
- Cohort 2: HIV infected subjects
  Interventions: Biological: 4CMenB (Bexsero®) vaccine
- Cohort 3: Patients candidates for / in treatment with biological drugs such as monoclonal antibodies anti CD-20 (rituximab or ocrelizumab)
  Interventions: Biological: 4CMenB (Bexsero®) vaccine

INTERVENTIONS:
Biological: 4CMenB (Bexsero®) vaccine — Participants will receive 2 doses of 4CMenB (Bexsero®) vaccine administered intramuscularly 1-2 months apart

SUMMARY:
The meningococcal quadrivalent conjugate vaccine (MenACWY) and the licenced multicomponent MenB vaccine (Bexsero®) have already been included in the Italian childhood immunization programme and recommendations for high risk categories have been also implemented.

As by NIP, vaccination against MenB with either 4CMenB or fHbp-MenB is offered for free for several conditions including subjects with severe primary or secondary immunodeficiency.

In Liguria Region meningococcal vaccination is actively offered to several chronic conditions including asplenia, patients with lymphoproliferative disease (also HSCT), subject treated with anti-CD20 mAb and HIV-positive.

In Liguria Region there is a large diverse population with risk condition that, as by national and regional recommendation, receive meningococcal vaccination. For some of them, i.e. asplenic and complement deficiencies groups, evidence have been generated through an ad hoc clinical trial, while for other important groups there is clear need of immunogenicity data.

In the proposed study, the Investigators plan to administer two doses of MenB vaccine (Bexsero®), 1-2 months apart, to adult patients living in Genoa area and belonging to following categories:

* Bone marrow transplant (HSCT patient)
* HIV positive
* Alfa-CD20 subjects (i.e. Patients candidates for / in treatment with biologic drugs such as Rituximab).

Immunogenicity data will be then obtained from sera collected at the day of the first Bexsero dose and one month after the immunization course by Serum Bactericidal Activity (SBA) assay.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 18 through 65 years of age at the time of enrollment who are high risk for IMD, including subjects with documented medical history of any of the following criteria:

  1. Hematopoietic Stem Celi Transplantation (allogenic or autologous stem celi transplant)
  2. HIV infection
  3. candidate for / in treatment (ongoing) with biological drugs such as monoclonal antibodies anti CD- 20 (rituximab or ocrelizumab)
* Written informed consent obtained from the subject (or legal representative).
* Subjects (or legal representative) who are able to comprehend all procedures and to comply with the study requirements

Exclusion Criteria:

* Subjects not able to understand and to adhere to ali study procedures
* Subjects aged <18 or >65 years
* Known or suspected allergy/hypersensitivity to any vaccine component
* History of serious adverse reaction to any vaccine
* Administration of immunoglobulins and/or any blood products within 3 months prior to enrollment or planned administration during the entire study period
* History of any meningococcal group B vaccination or having been diagnosed with meningococcal disease ever before
* Stem celi transplantation within 6 months before the enrollment to the study
* HIV-infected patients with detectable viral load (>50 copies/mL) and/or CD4 celi count < 200 cells/mm3 in the last 6 months
* Receipt of any vaccine within 28 (for live vaccines) or 14 (for no-live vaccines) days prior to study vaccination
* Planned vaccination (other than the study vaccination) during the entire study period
* Fever or any acute disease or infection within 3 days prior to vaccination
* Receipt of any antibiotics within 3 days before enrollment
* Coagulation disorder contraindicating intramuscular vaccination Any condition that in the opinion of the investigator would pose a health risk to the subject if enrolled or could interfere with the study procedures
* Current participation to another investigational study or planned enrollment to an investigational during the entire study period
* Planned surgery or hospitalization during the entire study period
* Subjects who participated in Cohort 1, 2 or 3, cannot be included in other different cohorts
* Pregnancy or breastfeeding (asking the woman to sign a declaration that she is not pregnant or breastfeeding).
* Any contraindication to the study vaccine (Bexsero®) as specified in the Summary of Product Characteristics.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects aged 18 to 65 years with an acquired immune deficiency, including three study groups:
  * Cohort l-Hematopoietic Stem Celi Transplant (HSCT) patients
  * Cohort 2-HIV infected subjects
  * Cohort 3-patients candidates for / in treatment with biological drugs such as monoclonal antibodies anti CD-20 (rituximab or ocrelizumab)
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2020-02-06 (Actual); Primary Completion 2024-01-11 (Actual); Study Completion 2024-01-11 (Actual)

PRIMARY OUTCOMES:
hSBA geometries mean titres (GMTs) against relevant MenB strains | baseline (Visit 1) and one month after the second vaccination (Visit3).
  hSBA geometries mean titres (GMTs) against relevant MenB strains
4 fold increase in hSBA against relevant MenB | Baseline to one month after the second vaccination (Visit3)
  The proportion of subjects with at least 4 fold increase in hSBA against relevant MenB strains from baseline to one month after the second vaccination (Visit3)
hSBA titres >1:4 against relevant MenB strains at Visit3 (one month after the second vaccination) | One month after the second vaccination (Visit3)
  The proportion of subjects with "protective" hSBA titres >1:4 against relevant MenB strains at Visit3 (one month after the second vaccination).

SECONDARY OUTCOMES:
Local and systemic AEs | 7 days (including the day of vaccination) after Visits 1 and 2.
  The incidence of subjects with solicited local and systemic AEs (Pain, Erythema, Swelling, Induration, Fever -body temperature ~38.0°C-, Nausea, Myalgia, Arthralgia, Headache, Fatigue) up to 7 days (including the day of vaccination) after Visits 1 and 2.
Unsolicited AEs | 7 days (including the day of vaccination) after Visits 1 and 2.
  The incidence of subjects with any other unsolicited AEs up to 7 days (including the day of vaccination) after Visits 1 and 2.
SAEs and AEs leading to withdrawal and medically attended visits throughout the study period | An average of 15 months (from the day of first vaccination to the end of the study)
  The incidence of subjects with SAEs and AEs leading to withdrawal and medically attended visits throughout the study period

CONTACTS AND LOCATIONS:
Locations (1):
- U.O.Igiene Ospedale Policlinico San Martino - IRCCS, Genoa, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Miller EC, Chase NM, Densen P, Hintermeyer MK, Casper JT, Atkinson JP. Autoantibody stabilization of the classical pathway C3 convertase leading to C3 deficiency and Neisserial sepsis: C4 nephritic factor revisited. Clin Immunol. 2012 Dec;145(3):241-50. doi: 10.1016/j.clim.2012.09.007. Epub 2012 Sep 28. PMID 23117396
- [Background] Salit IE. Meningococcemia caused by serogroup W135. Association with hypogammaglobulinemia. Arch Intern Med. 1981 Apr;141(5):664-5. PMID 6784688
- [Background] Miller L, Arakaki L, Ramautar A, Bodach S, Braunstein SL, Kennedy J, Steiner-Sichel L, Ngai S, Shepard C, Weiss D. Elevated risk for invasive meningococcal disease among persons with HIV. Ann Intern Med. 2014 Jan 7;160(1):30-7. doi: 10.7326/0003-4819-160-1-201401070-00731. PMID 24166695
- [Background] Abio A, Neal KR, Beck CR. An epidemiological review of changes in meningococcal biology during the last 100 years. Pathog Glob Health. 2013 Oct;107(7):373-80. doi: 10.1179/2047773213Y.0000000119. Epub 2013 Dec 19. PMID 24392681
- [Background] Cohn AC, MacNeil JR, Harrison LH, Hatcher C, Theodore J, Schmidt M, Pondo T, Arnold KE, Baumbach J, Bennett N, Craig AS, Farley M, Gershman K, Petit S, Lynfield R, Reingold A, Schaffner W, Shutt KA, Zell ER, Mayer LW, Clark T, Stephens D, Messonnier NE. Changes in Neisseria meningitidis disease epidemiology in the United States, 1998-2007: implications for prevention of meningococcal disease. Clin Infect Dis. 2010 Jan 15;50(2):184-91. doi: 10.1086/649209. PMID 20001736
- [Background] Crum-Cianflone N, Sullivan E. Meningococcal Vaccinations. Infect Dis Ther. 2016 Jun;5(2):89-112. doi: 10.1007/s40121-016-0107-0. Epub 2016 Apr 16. PMID 27086142
- [Background] Conferenza Stato-Regioni il 19 gennaio 2017. Piano Nazionale Prevenzione Vaccinale 2017-2019 (PNPV). Gazzetta Ufficiale del 18 febbraio 2017
- [Background] Regione Liguria DGR n. 284 del 07/04/2017. Piano Regionale in Prevenzione Vaccinaleaggiornamento 2017. http://www.alisa.liguria.it/index.php?option=com_docman&task=search_result&ltemi d=323.
- [Background] Martinon-Torres F, Bernatowska E, Shcherbina A, Esposito S, Szenborn L, Marti MC, Hughes S, Faust SN, Gonzalez-Granado LI, Yu LM, D'Agostino D, Calabresi M, Toneatto D, Snape MD. Meningococcal B Vaccine Immunogenicity in Children With Defects in Complement and Splenic Function. Pediatrics. 2018 Sep;142(3):e20174250. doi: 10.1542/peds.2017-4250. Epub 2018 Aug 1. PMID 30068713
- [Result] Ram S, Lewis LA, Rice PA. Infections of people with complement deficiencies and patients who have undergone splenectomy. Clin Microbiol Rev. 2010 Oct;23(4):740-80. doi: 10.1128/CMR.00048-09. PMID 20930072